CLINICAL TRIAL: NCT03326453
Title: Effect of Mini Implants Supported Over Dentures Versus Conventional Implant After Bone Expansion in Thin Mandibular Ridge on Patient Satisfaction:
Brief Title: Effect of Mini Implants Supported Over Dentures Versus Conventional Implant After Bone Expansion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Osama Ahmed Aboelfetooh, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-10-16
Record Dates: First submitted 2017-10-12; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Complete Edentulism
Keywords: mini dental implant; overdenture; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Dental Implants

STUDY DESIGN:
Who Masked: Participant
Masking Description: The Principal investigator ,main supervisor and co-supervisor cannot be blinded as the implant placement technique for both groups will be different. In addition during assessment of 2ry outcome (bone height change) the x-ray will reveal the difference in the shape of both types of implants thus assessor couldn't be blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mini Dental implant (Experimental): 2 mini dental implant of diameter 2.8 mm with length 10 mm will be inserted mandiblular ridge ≥5 mm mesial to the mental foraminato support overdentures for the intervention group.
  Interventions: Device: Mini dental implant
- conventional implant (No Intervention): two slandered implant diameter 3.7 mm and length 10 mm will be placed in interforaminal region of mandiblular ridge support overdenture for the compartor group.

INTERVENTIONS:
Device: Mini dental implant — titanium mini dental implant which diameter less than 3 mm
  Other Names: narrow dental implant
  Arms: Mini Dental implant

SUMMARY:
The better form of ridge will provide using wider implants that can have better abilities to with stand forces and to prevent alveolar bone loss as much as possible. Ridge expansion gained some popularity due to easiness compared to any other procedure that can gain bone. However, this treatment modality needs to be evaluated as compared to Mini Dental Implants (MDIs) over denture in thin mandibular ridge.

In mandibular edentulous patients having thin ridge, does the mini implant supported over denture, compared to the conventional implant supported over denture after bone expansion affect bone height around implants?

DETAILED DESCRIPTION:
PICO

P: Completely edentulous Patients.

I: Mandibular overdenture supported by mini dental implant.

C: Mandibular overdenture supported by conventional implant diameter after bone expansion.

O: outcomes as follows:

Primary Outcome: Patient satisfaction, Questionnaire Visual analog scale (VAS), Measuring unit: Mm. (Geckili et al.

Secondary Outcome: Bone height change, Measuring device: DIGORA® X ray, Measuring unit: Mm.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients ranging from age 35 to 75 years
* Angle's Class I skeletal relationship
* Normal facial symmetry
* Cooperative patients
* Adequate inter-arch space not less than 12mm

Exclusion Criteria:

* Temporomandibular disorders
* Uncontrolled diabetes
* Bleeding disorders or anticoagulant therapy
* Flabby tissues or sharp mandibular residual ridge.
* Heavy smokers.
* Patient's with neuromuscular disorders
* Patients on chemotherapy or radiotherapy
* Severe psychiatric disorders
* Angle's class II and III skeletal relationship

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
patients satisfaction | after six months of over denture insertion
  Visual analogue scale: a scale from 0-10 where 0 represents unsatisfied and 10 represents highly satisfied.

SECONDARY OUTCOMES:
Bone height change | baseline (T0) initial bone height (millimetres), after six months usage of over denture(T1) bone height (millimetres), then after twelve-months usage of over denture(T2) bone height. 1st period (T1-T0) after 6 months 2nd period (T2-T1) after 12 months
  measure the amount of bone height change in (millimetres) of all implant placed by DIGORA® X ray and Calliper device.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Souza RF, Ribeiro AB, Della Vecchia MP, Costa L, Cunha TR, Reis AC, Albuquerque RF Jr. Mini vs. Standard Implants for Mandibular Overdentures: A Randomized Trial. J Dent Res. 2015 Oct;94(10):1376-84. doi: 10.1177/0022034515601959. Epub 2015 Aug 20. PMID 26294416